CLINICAL TRIAL: NCT03857126
Title: Surveillance fœtale assistée Par Ordinateur - Obstétrique
Brief Title: Computer-assisted Fetal Monitoring - Obstetrics
Acronym: SURFAO-Obst
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other); University Grenoble Alps (Other); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Other Study IDs: 38RC18.172
Record Dates: First submitted 2018-12-31; First posted 2019-02-27 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: ECG-PCG-CTG Acquisition on Pregnant Voluntary Subjects
Keywords: Signal Database; Pregnancy; Electrocardiogram; Phonocardiogram; Cardiotocography; Usability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnancy volunteer subjects: Subjects who will agree to participate in the investigator's study will be pregnant healthy subjects with no particular antecedent, followed at the University Hospital of Grenoble for a physiological pregnancy; their child will be not affected by any prenatal pathology.
  Subjects will be enrolled in a 30 min monitoring phase to collect signals from ECG-PCG-CTG abdominal and thoracic non invasive sensors.
  Interventions: Other: Signal acquisition

INTERVENTIONS:
Other: Signal acquisition — ECG-PCG-CTG synchronized signals acquisition over a monitoring phase of 30 minutes. These signals will be acquired with passive non invasive sensors (abdominal and thoracic).
  Other Names: Non invasive ECG-PCG-CTG sensors

SUMMARY:
In the context of fetal heart monitoring, the SurFAO project offers an alternative to current clinical routines. The challenge is to extract, from few non-invasive sensors on the maternal abdomen, a fetal electrocardiogram (ECGf) of great quality allowing a clinical diagnosis (follow-up of the FHR (fetal heart rate)) and extraction of ECG waveforms).

The proposed approach proposes a technological breakthrough shared by a consortium of researchers and clinicians. The originality is driven by innovative methodological choices: the use of a multimodal system (ECG coupling with PCG (phonocardiographic)) for the signal acquisition in order to increase the robustness of information extraction, by taking into account clinical uses and the need for the monitoring process support, and by setting up a reference for this multimodal database.

The objective is to feed a database that will be used in the future to develop ECGf extraction methods estimating the FHR.

DETAILED DESCRIPTION:
To monitor the well-being of a fetus or for a clinical diagnosis, a challenge is to extract a fetal electrocardiogram (fECG) signal of high quality from a limited number of non-invasive sensors on the maternal abdomen.

During childbirth, fetal monitoring is assessed by the fetal heart rate (FHR), classically from cardiotocography (CTG). The aim is to monitor FHR variability anomalies that reflect a too high fetal malaise. It is very common to have difficulties to reliably record FHR due to confusion of rhythms of the mother and the fetus that can lead to unnecessary caesareans. With 800000 childbirths in France per year, improving the reliability of FHR estimation by fECG analysis is therefore of high clinicalinterest.

To deal with, the proposed approach aims at coupling two complementary cardiac information acquired at the best-located position. Therefore, the proposed solution is (i) to combine the use of electrophysiological sensors ECG and acoustic sensors of microphonic type that can register phonocardiographic signals (PCG), (ii) to assist by computer the clinical expertise to choose the best sensors location. Several methodological aspects will be considered: to improve the robustness of the FHR estimation with degraded signals based on multimodality, to overcome some practical limitations to extract the fECG waveforms by enhancing the process extraction with PCG and to assist the user in the sensors choice and placement by predicting their best locations and their kinds (ECG or PCG).

The SurFAO project proposes then an original approach of computer-assisted fetal monitoring and thus differs from previous published works of fECG extraction solutions, only based on algorithmic performances mostly in well-controlled situations. The original aspects of the investigator's proposal are the innovative methodological choices based on multimodality and informed recording process, the consideration of the medical uses and of the necessity to help the clinical monitoring to design the algorithms, the new reference multimodal database, and the academic-clinical consortium, that will guarantee the relevance of all proposed parts.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant of a single pregnancy,
* Aged over 18,
* During the 9th month of pregnancy (>= 37 weeks),
* With uncomplicated maternal and fetal pregnancy follow-up,
* With a BMI between 18.5 and 30 at the beginning of pregnancy,
* Without a notable medical history,
* Enrolled in a social security scheme,
* Having signed the consent form for the study.

Exclusion Criteria:

* Subject under guardianship, protected by law or deprived of liberty (Article L1121-8),
* Subject under administrative or judicial supervision,
* Subject in exclusion period of another study,
* With toxic consumption (i.e. tobacco, alcohol, cannabis),
* With inaccurate pregnancy term,
* With denial of pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
ECG Signals Database | 30 minutes
  Synchronized signals from ECG electrodes during a 30-minute monitoring phase. Tracking of the electrical activity in the heart. During the study period we will collect R wave, P wave, QT interval, ST interval, QRS complex, RR interval components of the ECG.
  Signals were then processed to extract fetal ECG.
PCG Signals Database | 30 minutes
  Synchronized signals from PCG sensors during a 30-minute monitoring phase. Acquisition of acoustic information reflecting the contraction and relaxation of the heart.
  During the study period we will collect S1 and S2 sounds components of the PCG. Signals were then processed to extract fetal PCG.
CTG Signals Database | 30 minutes
  CTG is continuous monitoring of the fetal heart rate (gold standard reference). Physicians evaluate specific clinical CTG parameters by means of visual inspection.

SECONDARY OUTCOMES:
Subject Acceptability: Score | 15 minutes
  The subject acceptability score will be composed by the addition of 7 scales. These scales have been specifically created for the SurFAO system. The score can go from 0 (worst) to 70 (best). Each scale can give from 0 to 10 points to the final score.
Subject Acceptability : Descriptive analysis | 15 minutes
  Open questions will be asked to the subjects in a questionnaire. A descriptive analysis will be done with the answers.
Use Error evaluation : System Usability Scale (SUS) | 15 minutes
  The System Usability Scale (SUS) is a validated tool for assessing the subjective usability of a system, in this case, the SurFAO System. It contains 10 questions that are rated on a scale from 1 to 5. "The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100." Jeff Sauro established the average score of SUS is 68.
  The score can go from 0 (worst) to 100 (best).
Use Error evaluation : Descriptive analysis | 15 minutes
  In a journal, the users will write their difficulties using the system. A descriptive analysis will be done with the answers.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Equy, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Equy V, Buisson S, Heinen M, Schaal J-P, Hoffmann P, Sergent F. Confusion between maternal and fetal heart rate during delivery: risk factors and consequences British Journal of Midwifery, vol.20 (11), 2012
- [Result] Gobillot S, Fontecave-Jallon J, Equy V, Rivet B, Gumery PY, Hoffmann P. Non-invasive fetal monitoring using electrocardiography and phonocardiography: A preliminary study. J Gynecol Obstet Hum Reprod. 2018 Nov;47(9):455-459. doi: 10.1016/j.jogoh.2018.08.009. Epub 2018 Aug 23. PMID 30144558
- [Result] Noorzadeh S, Rivet B, Gumery PY. An application of Gaussian processes on ocular artifact removal from EEG. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:554-7. doi: 10.1109/EMBC.2015.7318422. PMID 26736322
- [Result] Noorzadeh S, Niknazar M, Rivet B, Fontecave-Jallon J, Gumery PY, Jutten C. Modeling quasi-periodic signals by a non-parametric model: application on fetal ECG extraction. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1889-92. doi: 10.1109/EMBC.2014.6943979. PMID 25570347
- [Result] Noorzadeh S, Rivet B, Guméry PY. A multi-modal approach using a non-parametric model to extract fetal ECG. Proc. IEEE Int. Conf. Acoustics, Speech, and Signal Processing (ICASSP), Brisbane, Australia, 2015, pp. 1856-60